CLINICAL TRIAL: NCT03330691
Title: Pediatric and Young Adult Leukemia Adoptive Therapy (PLAT)-05: A Phase 1 Feasibility and Safety Study of Dual Specificity CD19 and CD22 CAR-T Cell Immunotherapy for CD19+CD22+ Leukemia
Brief Title: A Feasibility and Safety Study of Dual Specificity CD19 and CD22 CAR-T Cell Immunotherapy for CD19+CD22+ Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director, Seattle Children's Therapeutics, Seattle Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLAT-05
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Leukemia; Lymphoma
Keywords: CD19; CD22; CAR T-cell
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patient-derived CD19- and CD22 specific CAR v1 (Experimental): Patient-derived CD19-specific CAR also expressing an HER2t and CD22-specific CAR T-cells also expressing an EGFRt
  Interventions: Biological: Patient-derived CD19- and CD22 specific CAR
- Patient-derived CD19- and CD22 specific CAR v2 (Experimental): Patient-derived CD19-specific CAR also expressing an HER2t and CD22-specific CAR T-cells also expressing an EGFRt
  Interventions: Biological: Patient-derived CD19- and CD22 specific CAR

INTERVENTIONS:
Biological: Patient-derived CD19- and CD22 specific CAR — Patient-derived CD19-specific CAR also expressing an HER2t and CD22-specific CAR T-cells also expressing an EGFRt

SUMMARY:
Patients with relapsed or refractory leukemia often develop resistance to chemotherapy and some patients who relapse following CD19 directed therapy relapse with CD19 negative leukemia. For this reason, the investigators are attempting to use T-cells obtained directly from the patient, which can be genetically modified to express two chimeric antigen receptors (CARs). One is to recognize CD19 and the other is to recognize CD22, both of which are proteins expressed on the surface of the leukemic cell in patients with CD19+CD22+ leukemia. The CAR enables the T-cell to recognize and kill the leukemic cell through recognition of CD19 and CD22. This is a phase 1 study designed to determine the safety of the CAR+ T-cells and the feasibility of making enough to treat patients with CD19+CD22+ leukemia.

ELIGIBILITY:
Inclusion Criteria:

* First 2 subjects: male and female subjects age ≥18 and < 27 years (as of 2/16/18 the first 2 subjects were enrolled and treated); subsequent subjects <31 years.
* Diagnosis of CD19+22+ leukemia
* Disease status:

  * If post allogeneic HCT: Confirmed CD19+CD22+ leukemia recurrence defined as at least 0.01% disease following allogeneic HCT
  * If relapse/refractory status with no prior history of allogeneic HCT, one of the following:
  * Second or greater marrow relapse, with or without extramedullary disease
  * First marrow relapse at end of first month or re-induction with marrow having at least 0.01 % blasts by morphology and/or MPF
  * Primary refractory as defined as greater than 5% blasts by multi-parameter flow after at least 2 separate induction regimens.
  * Subject has indication for HCT but has been deemed ineligible, inclusive of persistent MRD prior to HCT
* Asymptomatic from CNS involvement, if present, and in the opinion of the Principal Investigator with a reasonable expectation that disease burden can be controlled in the interval between enrollment and T-cell infusion. Subjects with significant neurologic deterioration will not be eligible for T-cell infusion until stabilized.
* Free from active GVHD and off immunosuppressive GVHD therapy for 4 weeks prior to enrollment
* Lansky or Karnofsky performance score of at least 50
* Life expectancy of at least 8 weeks
* Recovered from acute toxic effects of all prior chemotherapy, immunotherapy, and radiotherapy
* At least 7 days post last chemotherapy administration (excluding intrathecal maintenance chemotherapy)
* At least 7 das post last systemic corticosteroids administration (unless physiologic replacement dosing)
* No prior genetically modified cell therapy that is still detectable or virotherapy
* Adequate organ function
* Adequate laboratory values
* Willing to participate in long-term follow-up for up to 15 years, if enrolled in the study and receive T cell infusion
* Patients of childbearing/fathering potential must agree to use highly effective contraception from the time of initial T cell infusion through 12 months following the last T cell infusion

Exclusion Criteria:

* Presence of active clinically significant CNS dysfunction
* Pregnant or breast-feeding
* Unable to tolerate apheresis procedure
* Presence of active malignancy other than CD19+CD22+ leukemia
* Presence of active severe infection
* Presence of any concurrent medical condition that, in the opinion of the Principal Investigator, would prevent the patient from undergoing protocol-specified therapy

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2035-03-03 (Estimated)

PRIMARY OUTCOMES:
The adverse events associated with one or multiple CAR T-cell product infusions will be assessed | 30 days
  Type, frequency, severity, and duration of adverse events will be summarized
The number of successfully and unsuccessfully manufactured and infused CAR T-cell products will be assessed | 28 days
  Proportion of products successfully manufactured and infused

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Annesley, MD, Study Chair — Seattle Children's Hospital
Locations (5):
- United States (4):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Seattle Children's Hospital, Seattle, Washington
- Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh N. Modified T cells as therapeutic agents. Hematology Am Soc Hematol Educ Program. 2021 Dec 10;2021(1):296-302. doi: 10.1182/hematology.2021000262. PMID 34889384
- [Derived] Johnson AJ, Wei J, Rosser JM, Kunkele A, Chang CA, Reid AN, Jensen MC. Rationally Designed Transgene-Encoded Cell-Surface Polypeptide Tag for Multiplexed Programming of CAR T-cell Synthetic Outputs. Cancer Immunol Res. 2021 Sep;9(9):1047-1060. doi: 10.1158/2326-6066.CIR-20-0470. Epub 2021 Jul 9. PMID 34244298